CLINICAL TRIAL: NCT01632293
Title: Evaluating Intervention Responsiveness in People With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00068596
Record Dates: First submitted 2012-06-28; First posted 2012-07-02 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- exercise (Experimental): Individuals with multiple sclerosis and age and gender matched healthy controls will participate in a supervised exercise program for 12 weeks.
  Interventions: Behavioral: progressive resistance training

INTERVENTIONS:
Behavioral: progressive resistance training — The exercise program uses guided progressive resistance training to provide an individualized program of strength training. The progressive resistance training intervention will consist of 12 weeks of guided resistance training twice weekly; in addition, subjects will be instructed to do one day of progressive resistance training at the home weekly.
  Other Names: strength; exercise training

SUMMARY:
The purpose is to see how multiple sclerosis (MS) is associated with strength and sensation using MRI, in persons with MS. The investigators will also see whether exercise can improve these symptoms for persons with MS.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic inflammatory disorder that damages myelin sheaths and axons in the brain and spinal cord. Within ten years of being diagnosed with MS, a majority of people will experience disability, most often walking impairments. The currently available pharmacologic treatments offer protection from new attacks but do not help with recovery; thus, in many cases the only hope for improvement, is through physical rehabilitation.

Rehabilitative interventions, such as progressive resistance training (PRT), have been shown to improve strength and sometimes walking in many individuals with MS. However, there are also many individuals who do not respond, which tends to be ignored in the literature. In addition, most intervention studies measure the primary impairment (e.g, strength) with little or no consideration for other impairments (e.g., sensory loss) and any effects on more complicated movements (e.g. standing, or changing direction). Since MS is so heterogeneous, it would be helpful to know which individuals are likely to benefit from rehabilitation.

Standard MS care uses MRI for diagnosis, identification of inflammatory lesions, and determination of treatment efficacy. Conventional rehabilitation relies on clinical judgment, rating scales and impairment measures to determine treatment efficacy. The investigators would like to understand how behavioral impairments and MRI findings relate to each other, and predict rehabilitation potential for people with MS. The investigators have previously shown that damage measured using tract specific MRI, specifically magnetization transfer (MTI) and diffusion tensor imaging (DTI), correlates with physical impairments in individuals with MS. Here the investigators propose to determine whether measures of clinical impairment and tract specific MRI can improve our ability to predict who will respond best to a PRT exercise intervention by improving functional movement. The investigators will perform a PRT intervention. The investigators will measure sensory and motor impairments and walking ability before and after the intervention. MRI will be done before treatment to assess the integrity of critical motor (corticospinal, CST) and sensory (dorsal column-medial lemniscus, DC-ML) tracts across the cervical spinal cord and brain. The investigators hypothesize that a combination of impairment measures and MRI measure will predict improvement in functional movement following three months of PRT.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of MS
* If on immunomodulatory therapy, subjects have to have been on that therapy for at least 6 months prior to the start of the study.
* Medically stable
* Able to follow complex directions as determined by a score of less than or equal to 1 on a subset of questions taken from the NIH Stroke scale
* Normal passive range of motion at the hips, knees, and ankles with minimum to no pain

Exclusion Criteria:

* Evidence of other neurological deficit that could interfere, such as previous stroke or muscle disease
* Congestive heart failure
* MS exacerbation within 8 weeks of study start
* MS exacerbation affecting CST or DC-ML tracts
* peripheral artery disease with claudication
* cancer
* pulmonary or renal failure
* unstable angina
* uncontrolled hypertension (greater than 190/110 mmHg)
* orthopedic or pain conditions
* history of kidney disease, due to potential of gadolinium reactions leading to nephrogenic systemic fibrosis (NSF)
* because pregnancy may change the MRI signals that we are studying, we have chosen not to enroll pregnant women in this study

Healthy controls have the same age and exclusion criteria as people with multiple sclerosis except that they must have normal neurological function

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change in maximal voluntary contraction of the hip flexors from baseline to end of training and to post-training | Participants are assessed at baseline (visit 1, enrollment), end of training (visit 2, week 12) and post-training (visit 3, week 24).
  Here, we will assess whether the degree of a person's white matter integrity (i.e. for tracts of interest as measured from MRI) predicts their ability to benefit from exercise. Our prediction is that those individuals with preserved white matter integrity will show the greatest improvement in hip flexor strength.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Zackowski, Ph.D., Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (1):
- Motion Analysis Lab, Baltimore, Maryland, United States

REFERENCES:
- See also: Related Info — http://www.kennedykrieger.org/research-training